CLINICAL TRIAL: NCT03418233
Title: Regeneration of Ischemic Damages in Cardiovascular System Using Wharton's Jelly as an Unlimited Source of Mesenchymal Stem Cells for Regenerative Medicine. Project of the National Centre for Research and Development (Poland) 'STRATEGMED II'. Randomized Clinical Trial to Evaluate the Regenerative Capacity of CardioCell in Patients With Chronic Ischaemic Heart Failure (CIHF)
Brief Title: Randomized Clinical Trial to Evaluate the Regenerative Capacity of CardioCell in Patients With Chronic Ischaemic Heart Failure (CIHF)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: John Paul II Hospital, Krakow (Other)
Collaborators: KCRI (Other); National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CardioCell in CIHF
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: The CIHF trial will enroll 105 patients with randomization into active and placebo therapy with 2:1 ratio.
  Additional 5-10 subjects meeting inclusion/exclusion criteria will receive, in a non-blinded fashion, labelled CardioCell to determine the early myocardial uptake and retention of IMP.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Data and Safety Monitoring Board (DSMB) will be blinded at project start, but may request unblinding if necessary to accommodate effective review of data.
  Other than the DSMB (if necessary), the only other "un-blinded parties", meaning that they will have knowledge as to the patient's treatment assignment, will be the PBTiK UJ CM employee who participates in randomization utilizing randomization lists and investigational medication preparation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Active Comparator): Patients randomized to the active treatment group: Transcoronary or trans-bypass graft administration of CardioCell consist 30 000 000 cells (suspended in 20 ml of 0.9% NaCl and 5% albumin) will be performed using a dedicated cell delivery catheter.
  The cell delivery catheter is a typical coronary balloon catheter that is CE marked (1.2x10 mm balloon, RX system) modified to include cell delivery perforations in the balloon section of the catheter. The cell delivery catheter has been demonstrated not to affect cell viability or other cell properties.
  Interventions: Drug: CardioCell
- Control Group (Placebo Comparator): Patients randomized to the placebo group will receive Placebos consist 0.9% NaCl and 5% albumin injections (in the same volumes as CardioCell) via the coronary arter(ies)/bypass grafts. The CardioCell and placebo are distributed encoded, in an indistinguishable form.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: CardioCell — Patients randomized to the active treatment group will receive transcoronary or trans-bypass graft administration of 30 000 000 cells (suspended in 20 ml of 0.9% NaCl and 5% albumin).
  Injection will be performed using a dedicated cell delivery catheter. The cell delivery catheter is a typical coronary balloon catheter that is CE marked (1.2x10 mm balloon, RX system) modified to include cell delivery perforations in the balloon section of the catheter. The cell delivery catheter has been demonstrated not to affect cell viability or other cell properties.
  Other Names: CardioCell administration
  Arms: Active Group
Drug: Placebos — Patients randomized to the placebo group will receive Placebos consist 0.9% NaCl and 5% albumin injections (in the same volumes as CardioCell) via the coronary arter(ies)/bypass grafts. The CardioCell and placebo are distributed encoded, in an indistinguishable form.
  Other Names: Placebo administration
  Arms: Control Group

SUMMARY:
The main objective of the CIRCULATE project is to compare the clinical outcomes of CardioCell administration in treatment of ischemic damages of cardiovascular system with control group, who will receive the placebo.

DETAILED DESCRIPTION:
The CIHF trial will enroll 105 patients with randomization into active and placebo therapy with 2:1 ratio.

Additional 5-10 subjects meeting inclusion/exclusion criteria will receive, in a non-blinded fashion, labelled CardioCell to determine the early myocardial uptake and retention of IMP.

The primary research question of this project is to check if the administration of CardioCell could improve the clinical outcomes in patients with CIHF. There are several secondary questions, defined by secondary endpoints in each cohort, e.g.: if the investigated treatment is possible to administered, if the investigated treatment and way of CardioCell administration is safe, if it is possible to define any selected subgroup in which the treatment results are significantly different than in whole group.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* Diagnosis of ischemic heart failure (supported by history of CAD or revascularization by PCI or CABG procedure) without known need for revascularization or feasibility of revascularization
* Substantial chronic ischemic myocardial injury as demonstrated by LVEF ≤45% by SPECT and the clinical stage of NYHA II or III
* At least 50% viable myocardium (SPECT)
* Patency of at least two major coronary arteries and/or bypass grafts supplying their territories (confirmed in angiography within 12 months)
* Clinically stable CIHF for at least 3 months on guideline recommended therapy
* Signed informed consent

Exclusion Criteria:

* Other than ischemic cause of cardiomyopathy
* Less than 3 months from any substantial therapeutic intervention (such as, e.g. CRT/ICD fitting or revascularization)
* Less than 3 months from ACS
* BMI lower than 18 or greater than 45kg/m2
* Severe valvular heart disease or left ventricle aneurysm requiring aneurysmectomy or other structural interventions
* Candidate for heart transplantation
* Active or any history of malignancy or tumor
* Moderate or severe immunodeficiency
* Chronic immunosuppressive therapy
* Acute or chronic infection
* Coagulopathies
* Known alcohol or drug dependence
* Severe renal dysfunction (eGFR<20mL/min)
* Soft tissue disease or local infection in a place of required artery puncture
* Pregnancy or breastfeeding
* Females of childbearing potential who do not use a highly effective method of contraception
* Females of childbearing potential in absence of a negative highly sensitive urine or serum pregnancy test
* Participation in any other clinical research study that has not reached the primary efficacy endpoint or otherwise would interfere with the patient's participation in this project
* Life expectancy < 12 months
* Any objective or subjective reason for inability to attend follow-up visits
* Any concurrent disease or condition that, in the opinion of the investigator, would make the patient unsuitable for participation in the project

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Left ventricle ejection fraction (LVEF) increase | 6 months FU
  Left ventricle ejection fraction (LVEF) increase, assessed by SPECT at 6M FU vs. during index (baseline) imaging - comparison between two groups (active vs placebo therapy).

SECONDARY OUTCOMES:
An increase the result of 6 minute walk test | 3 and 6 month FU
  An increase the result of 6 minute walk test at 3 and 6 month.
Myocardial perfusion improvement | 6 month FU
  Myocardial perfusion improvement assessed in SPECT at 6 month FU.
Myocardial perfusion improvement | 6 month FU
  Myocardial perfusion improvement assessed in cardiac MRI at 6 month FU.
An improvement the result of spiroergometric test | 6 month FU
  An improvement the result of spiroergometric test at 6 month FU.
Left ventricle ejection fraction (LVEF) change against baseline | 6 month FU
  Left ventricle ejection fraction (LVEF) change (in %) against baseline, assessed in echocardiography.
Left ventricle end-systolic volume (ESV) change against baseline | 6 month FU
  Left ventricle end-systolic volume (ESV, in ml) change against baseline, assessed in echocardiography.
Left ventricle end-diastolic volume (EDV) change against baseline | 6 month FU
  Left ventricle end-diastolic volume (EDV, in ml) change against baseline, assessed in echocardiography.
NT pro-BNP level | 3, 6 and 12 months FU
  NT pro-BNP level at 3, 6 and 12 months in comparison to the baseline level.
The occurrence of major adverse cardiovascular events | 6 month and 1 year FU
  The occurrence of major adverse cardiovascular events (MACE including death, myocardial infarction, and hospitalization for heart failure) at 6 month and 1 year FU.
Quality of life improvement | 6 month and 1 year FU
  Quality of life improvement, assessed by SF-36 questionnaire or other dedicated for investigated population at 6 month and 1 year FU.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Musiałek, MD, PhD, Principal Investigator — John Paul II Hospital
Locations (5):
- Poland (5):
  - Instytut Kardiologii im. Prymasa Tysiąclecia Stefana Kardynała Wyszyńskiego, Katowice
  - Leszek Giec Upper-Silesian Medical Centre of the Silesian Medical University in Katowice, Katowice
  - The John Paul II Hospital, Krakow
  - The University Hospital in Cracow, Krakow
  - Central Clinical Hospital of the MSWiA in Warsaw, Warsaw